CLINICAL TRIAL: NCT05933031
Title: A Randomized, Double-Blind, Active-controlled, Multi-center, Therapeutic Exploratory Study to Evaluate the Safety and Efficacy of a Standard Triple Therapy With Tegoprazan (by Dose) in H. Pylori Positive Patients
Brief Title: Exploratory Study to Standard Triple Therapy With Tegoprazan(by Dose) in H. Pylori Positive Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IN_APA_E02
Record Dates: First submitted 2023-05-23; First posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Helicobacter Pylori Infection
MeSH Terms: interventions — tegoprazan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tegoprazan 50 mg (Experimental): Tegoprazan 50 mg/Clarithromycin/ Amoxicillin BID peroral, 14 days
  Interventions: Drug: Tegoprazan 50 mg Triple Therapy
- Tegoprazan 100 mg (Experimental): Tegoprazan 100 mg/Clarithromycin/ Amoxicillin BID peroral, 14 days
  Interventions: Drug: Tegoprazan 100 mg Triple Therapy
- Lansoprazole (Active Comparator): Lansoprazolee/Clarithromycin/ Amoxicillin BID peroral, 14 days
  Interventions: Drug: Lansoprazole Triple Therapy

INTERVENTIONS:
Drug: Tegoprazan 50 mg Triple Therapy — Tegoprazan 50 mg/Clarithromycin/ Amoxicillin BID peroral, 14 days
  Arms: Tegoprazan 50 mg
Drug: Tegoprazan 100 mg Triple Therapy — Tegoprazan 100 mg/Clarithromycin/ Amoxicillin BID peroral, 14 days
  Arms: Tegoprazan 100 mg
Drug: Lansoprazole Triple Therapy — Lansoprazole/Clarithromycin/ Amoxicillin BID peroral, 14 days
  Arms: Lansoprazole

SUMMARY:
This exploratory study is designed to compare safety and efficacy between a Tegoprazan dose-specific standard triple therapy and Lansoprazole standard triple therapy in H. pylori positive patients.

DETAILED DESCRIPTION:
A Randomized, Double-Blind, Active-controlled, Multicenter, Therapeutic Exploratory Study to to Evaluate the Safety and Efficacy of a Standard Triple Therapy with Tegoprazan and Lansoprazole standard triple therapy in H. pylori Positive Patients, twice a day for 14 days.

ELIGIBILITY:
Inclusion Criteria:

* H. pylori positive at screening
* Subjects who have upper gastrointestinal disease

Exclusion Criteria:

* Having received prior therapy for eradication of H. pylori
* Prior use of P-CAB, proton pump inhibitors (PPIs), H2 receptor blockers within 14 days
* Prior use of H. pylori eradication effective antibiotics, bismuth within 28 days

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 381 (Estimated)
Dates: Start 2023-02-27 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
H. pylori eradication rate | 42 days
  Assess H. pylori eradication rate by UBT

CONTACTS AND LOCATIONS:
Overall Officials: Jae Gyu Kim, Principal Investigator — Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Locations (1):
- Chung-Ang University Hosptial, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park JY, Hong SJ, Choi IJ, Baik GH, Kim SM, Park JJ, Jeon SW, Kim KO, Lee SK, Jung HY, Oh JH, Park CH, Kim SW, Shim KN, Jee SR, Moon HS, Moon JS, Choi CW, Lee WS, Kim JG. Tegoprazan-Based Triple Therapy for Helicobacter pylori Eradication: A Phase III Multicenter Randomized Clinical Trial. Helicobacter. 2026 Jan-Feb;31(1):e70106. doi: 10.1111/hel.70106. PMID 41531249